CLINICAL TRIAL: NCT02753998
Title: Paclitaxel-coated Balloon Angioplasty Versus Standard Angioplasty for the Treatment of Stenosis of Arteriovenous Fistula
Acronym: ABISS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Bard Peripheral Vascular, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P150908
Record Dates: First submitted 2016-04-25; First posted 2016-04-28 (Estimated); Last update posted 2022-03-22 (Actual); Status verified 2022-03

CONDITIONS: Angioplasty; Stenosis of Arteriovenous Fistula
Keywords: Stenosis of arteriovenous fistula; Angioplasty; Paclitaxel-Coated Balloon Angioplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional angioplasty + paclitaxel-coated balloon (Experimental): Treatment of stenosis of AVF by conventional angioplasty + 1 minute additional angioplasty with paclitaxel-coated balloon
  Interventions: Combination Product: Additional angioplasty with paclitaxel-coated balloon; Procedure: Conventional angioplasty
- Conventional angioplasty + placebo balloon (Placebo Comparator): Treatment of stenosis of AVF by conventional angioplasty + 1 minute additional angioplasty with placebo balloon.
  Interventions: Combination Product: Additional angioplasty with placebo balloon; Procedure: Conventional angioplasty

INTERVENTIONS:
Combination Product: Additional angioplasty with paclitaxel-coated balloon — Additional angioplasty with paclitaxel-coated balloon after conventional angioplasty
  Other Names: Lutonix® 035 balloon
  Arms: Conventional angioplasty + paclitaxel-coated balloon
Combination Product: Additional angioplasty with placebo balloon — Additional angioplasty with placebo balloon after conventional angioplasty
  Other Names: ClearPAC Omega® balloon
  Arms: Conventional angioplasty + placebo balloon
Procedure: Conventional angioplasty

SUMMARY:
The primary objective of this double-blind study is to compare the frequency of primary patency at 6 months in patients with stenosis of arteriovenous fistula (AVF) treated either by conventional angioplasty + angioplasty with balloon impregnated with paclitaxel or by conventional angioplasty + angioplasty with placebo balloon (balloon not impregnated with paclitaxel).

The other objectives of the study are:

1. To compare the frequency of primary patency at 3 months and 12 months.
2. To compare the rate of restenosis > 50% at the site of angioplasty at 3, 6 and 12 months.
3. To compare, at 3, 6 and 12 months, the proportion of patients with arteriovenous fistula deteriorating back to preoperative flow rate (within 20% of preoperative flow rate).
4. To compare, at 3, 6 and 12 months, the proportion of AVF with a flow rate < 500 ml / min.
5. To compare, at 3, 6 and 12 months, the cumulative rate of thrombosis.
6. To compare, at 3, 6 and 12 months, the medical costs related to direct medical care, initial treatments, monitoring, diagnosis and treatments of complications.

DETAILED DESCRIPTION:
Experimental design: prospective randomized, double blind, multicenter controlled study, with 2 experimental arms.

12 centers will participate in France, targeting to enrol 150 patients in total. Each patient will undergo angiography at the beginning of the intervention in order to confirm the presence of only one stenosis, to assess the degree of stenosis and to evaluate the vascular diameter.

All patients will first undergo angioplasty using standard balloons. thereafter, depending on randomization arm, an additional angioplasty will be performed during 1 minute with a paclitaxel impregnated balloon (active arm) or with a placebo balloon (placebo arm).

The duration of inclusion is planned for 18 months.

Each patient will have a 12-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years, man or woman.
* Chronic Hemodialysis.
* Native autologous arteriovenous fistula (AVF).
* AVF used at least once for hemodialysis.
* Preoperative flow measurement of AVF performed by Doppler.
* Length of the stenosis <120 mm.
* Outer diameter of the target vein <12mm.
* Hemodynamically significant Stenosis on AV fistula, defined according to international recommendations with the following two criteria:

  1. stenosis> 50% by Doppler or angiography,
  2. presenting at least one of the following :

     1. increased venous pressure during dialysis (venous pressure > 150 mmHg when blood flow measured at 200-225 ml / min, or venous pressure > 230 mmHg when blood flow measured at 400 ml / min);
     2. disappearance of thrill of AV fistula;
     3. increasing hemostasis time at the end of dialysis (> 20 minutes or increase by >=50% from usual hemostasis time);
     4. recirculation rate > 20%;
     5. flow of AVF < 500 ml / min responsible for a reduction of the flow of the dialysis circuit.
* Only one stenosis with significant impact hemodynamically.
* Signed informed consent.
* Patient has a health insurance.

Exclusion Criteria:

* Pregnant or breastfeeding women.
* Severe allergy to iodinated contrast agents, or to heparin, or to paclitaxel.
* Anastomotic stenosis involving the afferent artery.
* Multiple hemodynamically significant stenoses.
* Hemodynamically significant central venous stenosis.
* Stent already in place in treated vascular site.
* Diameter of the vein immediately upstream of stenosis greater than the maximum diameter of active balloon.
* AVF in lower limb.
* Coagulation disorder (outside of VKA use).
* Active infection.
* Inability to comply with the protocol requirements.
* Life expectancy less than 1 year due to progressive disease (neoplasia, severe organ failure).
* Follow-up expected to be difficult.
* Patient under guardianship.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2022-02 (Actual); Study Completion 2022-03 (Actual)

PRIMARY OUTCOMES:
Cumulated incidence of loss of primary patency of AVF | At 6 months
  Double-blind comparison of cumulated incidence of primary patency at 6 months after treatment of stenosis of AVF by conventional angioplasty + additional angioplasty.
  Cumulated incidence of primary patency loss of AVF at 6 months post procedure.

SECONDARY OUTCOMES:
Cumulated incidence of primary patency loss of the target lesion | At 3 months and 12 months
  Comparison between arms of cumulated incidence of primary patency loss of treated lesion at 3 and 12 months after treatment of stenosis.
  By cumulated incidence with no need for target lesion revascularization.
Cumulated incidence of restenosis > 50% at the site of angioplasty | At 3, 6 and 12 months
  Comparison between the arms of cumulated incidence of restenosis > 50% at the site of angioplasty of treated lesion of AVF, by cumulated incidence with at least one restenosis at angioplasty site at 3, 6 and 12 months.
Cumulated incidence of deteriorating flow rate | At 3, 6 and 12 months
  Cumulated incidence at 3, 6 and 12 months of deteriorating back to preoperative flow rate of AVF: defined by the difference of flow rate < 20% between preoperative measurement and follow-up measurement.
  Incidence of back to preoperative flow rate will be cumulated.
Cumulated incidence of patients with a flow rate < 500 ml / min | At 3, 6 and 12 months
  Comparison between the arms of cumulated incidence with a flow rate < 500 ml/min after treatments of stenosis.
Cumulative rate of thrombosis | At 3, 6 and 12 months
  Comparison between the arms at 3, 6 and 12 months cumulative rate of thrombosis, by the proportion of thrombosis of AVF, number of restenosis and number of thrombosis.
Time period before event's appearance | At 12 months
  Comparison between the arms time periods before the events' appearance: restenosis at the same site, stenosis at another site, thrombosis of AVF, death.
Cumulated incidence of adverse event (AE) | At 12 months
  Comparison between the arms post procedure AE, by cumulated incidences of AE in 12 months post procedure.
Medical costs | At 3, 6 and 12 months
  Comparison between the arms at 3, 6 and 12 months the costs of treatments of AVF, by direct medical care, initial treatments, monitoring, diagnosis and treatment of complications.
Cumulative incidence of cardiovascular serious adverse event (SAE) | At 12 months
  Comparison between the arms at 12 months the cumulative incidence of cardiovascular SAE.
Cumulative incidence of death | At 12 months
  Comparison between the arms at 12 months the cumulative incidence of death.

CONTACTS AND LOCATIONS:
Overall Officials: Raphaël Coscas, MD, PhD, Principal Investigator — Service chirurgie vasculaire, Hôpital Ambroise Paré
Locations (1):
- Service chirurgie vasculaire, Hôpital Ambroise Paré, Boulogne-Billancourt, Hauts-de-Seine, France

IPD SHARING:
Plan to Share IPD: No